CLINICAL TRIAL: NCT05717036
Title: Refractix DSP and TS Meter-DSP Measurement Comparison
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Reichert, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13910000-TPR-30
Record Dates: First submitted 2023-01-11; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: serum total protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TS Meter-DSP Measurement and Refractix DSP Measurement: The study will involve blood serum samples from (36) participants. Participants will be those presenting at a plasma collection center for routine plasma donation. Ordinary pre-screening for plasma donation includes a fingerstick and the collection of one small capillary tube (<0.085ml) of blood. Participants will be asked to provide a second capillary tube (<0.085ml) of blood from this fingerstick.
  Interventions: Device: Serum Total Protein Measurement with TS Meter-DSP and Refractix DSP

INTERVENTIONS:
Device: Serum Total Protein Measurement with TS Meter-DSP and Refractix DSP — The two blood samples will be centrifuged and hematocrit measured per the plasma center's standard operating procedures. One participant sample will be dispensed onto the cleared TS Meter-DSP for a serum total protein measurement. This measurement will be used, along with other pre-screening information, to determine if the participant can donate plasma. The second participant sample will be dispensed onto the investigational Refractix DSP for a serum total protein measurement. It will be compared to the sample measurement taken on the cleared TS Meter-DSP.

SUMMARY:
The goal of this clinical trial is to compare the serum plasma measurement results between the FDA cleared TS Meter-DSP and investigational Refractix DSP. Study participants will be individuals being screened for plasma donation in a plasmaphereris center. The main question the study aims to answer is whether the measurement taken on the investigational Refractix DSP device is equivalent, defined as within +/- 0.3g/100ml, of the measurement taken on the TS Meter-DSP. Participants will be asked to provide a second capillary tube of blood (<0.085ml) from the fingerstick that is part of their routine pre-screening for plasma donation.

DETAILED DESCRIPTION:
The TS Meter-DSP and investigational Refractix DSP are digital refractometers intended for the quantitative measurement of total protein in human serum or plasma. The devices are intended for use in plasma collection centers and are not for diagnostic purposes. Serum/plasma samples are taken from a successful microhematocrit assay and dispensed via pipette on to the instruments. The instruments measure the temperature compensated refractive index of the serum or plasma sample and digitally convert refractive index to an accurate total protein value. Potential donors with a total protein level of between 6.0 g/100ml and 9.0 g/100ml and that meet other pre-screening requirements are permitted to donate plasma.

These devices are FDA Class I in vitro diagnostic devices; FDA Regulation Number 862.2800 Refractometer for clinical use; with Product Code PSM, Refractometer for Donor Testing.

Participants will be those presenting for plasma donation. Ordinary pre-screening for plasma donation includes a fingerstick and the collection of one small capillary tube (<0.085ml) of blood. Participants who have consented to this study will be asked to supply a second capillary tube (<0.085ml) of blood for the clinical trial. The two samples will be centrifuged and hematocrit measured per the plasma center's standard operating procedures. One sample will be dispensed onto the TS Meter-DSP for total protein measurement. This measurement will be used to determine the individual's eligibility to donate plasma. The second sample will be dispensed on to the investigational Refractix DSP for total protein measurement. The measurements from both devices will be recorded on the Case Report Form. The study requires (36) participants with total protein measurements between 6.0 g/100ml and 9.0 g/100ml.

The primary analysis of data will include:

1. a Grubb's test for outlying paired difference values will be performed. If outliers are detected and a plausible non-device failure mechanism can be identified (eg, operator or data entry error), the values will be excluded from the acceptance criterion calculations;
2. an alpha=0.05 level equivalence test with an equivalence interval of +/- 0.3 g/100ml will be performed using the TOST (Two One Sample Test) procedure. A paired t-test 90% confidence interval for the difference in paired sample measurements will be constructed and reported; and
3. calculate the percentage of measurement pairs falling outside of the +/-0.3 tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18 and 90 years old
* Subjects must be able and willing to provide signed informed consent
* Subjects must be able to follow study instructions

Exclusion Criteria:

* Insufficient amount of plasma sample for use on either device in the study.
* Plasma samples of with total protein measurements outside of the 6.0 g/100ml to 9.0 g/100ml range will be excluded from the data analysis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be individuals presenting at a plasma collection center for plasma donation.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-02-13 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Serum Total Protein Measurement Comparison | Samples will be collected over one or two days at the plasma center. Data analysis by sponsor will be completed within 8 weeks.
  The purpose of this study is to show the investigational Refractix DSP refractometer yields equivalent measurement results to the predicate device TS Meter-DSP through comparison testing using human plasma samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Hemarus Plasma, Lauderhill, Florida, United States

IPD SHARING:
Plan to Share IPD: No